CLINICAL TRIAL: NCT03111823
Title: Feasibility of a 6-Week Aerobic Exercise Program During Chemotherapy for Metastatic Colorectal Cancer
Brief Title: Exercise Program During Chemotherapy in Metastatic Colorectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3C-16-1; NCI-2016-01089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-16-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2017-04-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Stage IV Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (aerobic exercise) (Experimental): Patients undergo aerobic exercise sessions consisting of cycling or walking at a low-moderate intensity and progressing to moderate intensity for 30 minutes 2 times a week for up to 8 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo aerobic exercise sessions
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well aerobic exercise works in improving quality of life and health-related outcomes in patients with stage IV colorectal cancer undergoing chemotherapy. Aerobic exercise during chemotherapy may improve quality of life and reduce fatigue and inflammation in the blood related to heart disease and diabetes in patients with stage IV colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether a 6-week indoor or outdoor aerobic exercise program is feasible in patients with metastatic colorectal cancer (mCRC) undergoing chemotherapy and to explore patient's preferences for indoor versus (vs.) outdoor exercise.

II. To determine the effects of a 6-week indoor or outdoor aerobic exercise program on cancer-related fatigue and quality of life (QOL) in patients with mCRC.

SECONDARY OBJECTIVES:

I. To determine the effects of a 6-week indoor or outdoor aerobic exercise program on body composition (lean body mass, fat mass, body fat percentage [%]) and biomarkers of systemic inflammation (interleukin-6 [IL-6], tumor necrosis factor alpha [TNF-a], C-reactive protein [CRP]) in patients with mCRC.

TERTIARY OBJECTIVES:

I. To determine the effects of a 6-week exercise program on cardiovascular (CV) function.

OUTLINE:

Patients undergo aerobic exercise sessions consisting of cycling or walking at a low-moderate intensity and progressing to moderate intensity for 30 minutes 2 times a week for up to 8 weeks.

After completion of study treatment, patients are followed up for 6 weeks and at weeks 13, 19, and 31.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic (stage IV) colorectal cancer
* Undergoing chemotherapy (have had 1 or 2 chemotherapy cycles infused at time of data collection; this will allow for any systemic inflammatory changes due to chemotherapy to set in); only patients with 1st or 2nd line therapy will be included
* Able to initiate a supervised exercise program (free from any CV, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity)
* Free from uncontrolled chronic disease including diabetes, hypertension, or thyroid disease
* Currently participate in less than 60 minutes of physical activity/week
* Willing to travel to the exercise facility at University of Southern California (USC) (parking fees and public transportation permits will be provided)
* Speak English or Spanish

Exclusion Criteria:

* Uncontrolled hypertension or other uncontrolled chronic disease (e.g. diabetes mellitus, thyroid disease, pulmonary disease, etc)
* Moderate to highly active level of physical activity (e.g. currently participating in > 60 minutes of moderate aerobic activity weekly)
* Orthopedic or other restrictions or contraindications to exercise
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Total number of minutes exercised per week with >80% total weekly minutes (48/60 minutes) completed | Up to 6 weeks
  The study will assess the feasibility using average weekly minutes of exercise completion (minutes/week) of all participants. Feasibility will be determined based on the total number of minutes exercised per week with >80% total weekly minutes (48/60 minutes) completed deeming this trial as feasible.

SECONDARY OUTCOMES:
Change in biomarkers of systemic inflammation | Baseline up to 31 weeks
  Change in biomarkers will be examined by a paired sample t-test, with a level of significance set at p <0.05.
Change in cancer-related fatigue | Baseline up to 31 weeks
  Assessed by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale
Change in QOL | Baseline up to 31 weeks
  Assessed by the Functional Assessment of Cancer Therapy-Colorectal cancer (FACT-C)

OTHER OUTCOMES:
Change in arterial stiffness/geometry | Baseline up to 31 weeks
  Assessed by ultrasound
Change in endothelial function | Baseline up to 31 weeks
  Assessed by flow-mediated dilation

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Ph.D., Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California